CLINICAL TRIAL: NCT07182916
Title: Factors Associated With Early Readmission in Critical Care
Acronym: FRASC
Status: Not yet recruiting | Type: Observational
Sponsor: Société Française d'Anesthésie et de Réanimation (Other)
Responsible Party: Sponsor
Other Study IDs: FRASC / 2025-08
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Early Readmission to the ICU

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention /Observation: No intervention: observation of patients with early eeadmission to the ICU
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Only observation

SUMMARY:
The COVID-19 health crisis has highlighted pre-existing challenges in patient flow management within healthcare facilities, especially in critical care units. This has sparked debate regarding the sufficiency of critical care beds in France, while drawing attention to the lack of downstream structures. Inefficient patient flow, leading to bed occupancy bottlenecks, has been correlated with both critical care length of stay and morbidity. Unplanned early readmission to critical care further exacerbates these strains and prolongs hospital length of stay. Currently, no standardized criteria are available to guide safe discharge from critical care. A recent Delphi consensus study proposed a set of criteria, although largely subjective. The primary outcome of the present study is to identify factors associated with unplanned early readmission to critical care within 48 hours of discharge. Delayed discharge from critical care represents another major bottleneck contributing to system strain. The secondary outcome of this study is therefore to assess the proportion of critical care beds occupied by patients deemed ready for discharge by the medical team, as well as to analyze the reasons underlying such delayed transfers.

DETAILED DESCRIPTION:
The COVID-19 health crisis has highlighted pre-existing challenges in patient flow management within healthcare facilities, especially in critical care units. This has sparked debate regarding the sufficiency of critical care beds in France, while drawing attention to the lack of downstream structures. Inefficient patient flow, leading to bed occupancy bottlenecks, has been correlated with both critical care length of stay and morbidity. Unplanned early readmission to critical care further exacerbates these strains and prolongs hospital length of stay. Currently, no standardized criteria are available to guide safe discharge from critical care. A recent Delphi consensus study proposed a set of criteria, although largely subjective. The primary outcome of the present study is to identify factors associated with unplanned early readmission to critical care within 48 hours of discharge. Delayed discharge from critical care represents another major bottleneck contributing to system strain. The secondary outcome of this study is therefore to assess the proportion of critical care beds occupied by patients deemed ready for discharge by the medical team, as well as to analyze the reasons underlying such delayed transfers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Hospitalized or admitted to the ICU

Exclusion Criteria:

* Objection to the use of their data (by patient or a relative when applicable)
* Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged 18 years or older admitted to the ICU
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Early Readmission to the ICU | From the first day of recruitment to 48 hours after the end of recruitment
  Patients readmitted to the ICU less than 48 hours after their first discharge

SECONDARY OUTCOMES:
Readmission to the ICU | From the first day of admission to 30 days of follow up
  Patients readmitted to the ICU less than 30 days after their first discharge
30-days mortality | From the first day of admission to 30 days of follow up
  Patients dead by day 30 of the follow-up
Rate of bed occupancy by patients deemed fit for discharged | From the first day of the study to the 7th day of the study
  Patients still hospitalized in the ICU the day after they were deemed fit for discharge by the medical team

CONTACTS AND LOCATIONS:
Overall Officials: François DEPRET, Study Chair — Hôpital Saint-Louis, AP-HP

IPD SHARING:
Plan to Share IPD: Undecided